CLINICAL TRIAL: NCT06742502
Title: A Phase II, Multicenter Clinical Study of Sintilimab Combined With Rituximab Followed by R-CHOP Regimen in Patients With Previously Untreated Primary Mediastinal Diffuse Large B-Cell Lymphoma
Brief Title: Sintilimab Plus Rituximab Followed by R-CHOP Regimen in Untreated PMBL
Acronym: Si-Ri
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huiqiang Huang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Si-Ri
Record Dates: First submitted 2024-12-07; First posted 2024-12-19 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Primary Mediastinal Diffuse Large B-cell Lymphoma
Keywords: primary mediastinal diffuse large B-cell lymphoma; PD-1 antibody; R-CHOP
MeSH Terms: interventions — Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sintilimab plus rituximab followed by R-CHOP regimen (Experimental): Participants will first receive sintilimab plus rituximab for 2 cycles, followed by interim PET-CT assessments. If patients achieve CR or CMR, they will continue to receive 2 courses of sintilimab plus rituximab, followed by 4 cycles of R-CHOP. Patients will receive 6 courses of R-CHOP if they do not achieve CR or CMR after 2 cycles of sintilimab plus rituximab. Patients will undergo PET-CT assessment and will receive 6 cycles of maintenance treatment with nintedanib if CR/CMR/PR is achieved and will be withdrawn from the study if SD/PD occurs. Total treatment cycles will not exceed 14 cycles.
  Interventions: Drug: Sintlimab+Rituximab follwed by R-CHOP(Cyclophosphamide, doxorubicin, vincristine, prednisone)

INTERVENTIONS:
Drug: Sintlimab+Rituximab follwed by R-CHOP(Cyclophosphamide, doxorubicin, vincristine, prednisone) — First strategy of targeted immunotherapy followed by chemotherapy for PMBL. Participants will first receive sintilimab(200mg) plus rituximab(375mg/m2) for 2 cycles. If patients achieve CR or CMR, they will continue to receive 2 courses of sintilimab plus rituximab, followed by 4 cycles of R-CHOP. Patients will receive 6 courses of R-CHOP if they do not achieve CR or CMR after 2 cycles of sintilimab plus rituximab. Patients will undergo PET-CT assessment and will receive 6 cycles of maintenance treatment with nintedanib if CR/CMR/PR is achieved and will be withdrawn from the study if SD/PD occurs. Total treatment cycles will not exceed 14 cycles.
  Other Names: CD20 antibody plus PD-1 antibody followed by R-CHOP

SUMMARY:
The goal of this clinical study is to evaluate the efficacy and safety of sintilimab combined with rituximab followed by R-CHOP regimen in treatment-naïve patients with primary mediastinal diffuse large B-cell lymphoma. The main questions it aims to answer are:

1. Objective response rate of sintilimab combined with rituximab
2. Objective response rate after R-CHOP regimen

DETAILED DESCRIPTION:
Participants will first receive sintilimab plus rituximab for 2 cycles, followed by interim PET-CT assessments. If patients achieve CR or CMR, they will continue to receive 2 courses of sintilimab plus rituximab, followed by 4 cycles of R-CHOP. Patients will receive 6 courses of R-CHOP if they do not achieve CR or CMR after 2 cycles of sintilimab plus rituximab. Patients will undergo PET-CT assessment and will receive 6 cycles of maintenance treatment with nintedanib if CR/CMR/PR is achieved and will be withdrawn from the study if SD/PD occurs. Total treatment cycles will not exceed 14 cycles

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in clinical study and fully understand, informed consent and sign informed consent form (ICF);
2. Age ≥ 18 years and ≤ 75 years at the time of signing the ICF.
3. treatment-naïve, no anti-lymphoma therapy.
4. Primary mediastinal DLBCL was confirmed histopathologically at the study site.
5. Lugano clinical stage I-IV.
6. International Prognostic Score (IPI) 0-5.
7. Available tumor tissue samples obtained by previous or fresh core needle aspiration or resection.
8. ECOG score of 0-2.
9. Expected survival greater than 12 months.
10. Must have at least 1 evaluable or measurable lesion that meets the LYRIC 2016 response evaluation criteria for malignant lymphoma.
11. Adequate organ and bone marrow function, no severe hematopoietic dysfunction and heart, lung, liver, kidney, thyroid dysfunction and immunodeficiency.
12. Pulse oximetry values > 92% at rest.
13. Women of childbearing potential (WOBCP) must have a negative serum pregnancy test within 7 days before the first dose; WOBCP or men and their WOBCP partners should agree to use effective contraception from signing the ICF until 6 months after the last dose of study drug.

Exclusion Criteria:

1. Primary central nervous system lymphoma or secondary central nervous system involvement.
2. previous treatment with immune checkpoint inhibitors (PD-1, PD-L1, CTLA-4, etc.).

3 History of severe allergic or allergic reactions to humanized or murine monoclonal antibodies.

4. Patients with active autoimmune diseases that require systemic treatment within the past two years; patients with autoimmune diseases that do not require systemic treatment within the past two years may be enrolled.

5. Subjects requiring systemic glucocorticoid therapy or other immunosuppressive therapy for a condition within 14 days prior to starting study treatment [subjects are allowed to be treated with topical, ocular, intra-articular, intranasal, and inhaled glucocorticoids (with minimal systemic absorption); short-term (≤ 7 days) glucocorticoid prophylaxis (e.g., contrast agent allergy) or for the treatment of non-autoimmune diseases (e.g., delayed hypersensitivity due to contact allergens) is allowed]. Low dose steroid debulking therapy for large tumor burden may be excluded (prednisone 30 mg bid × 5 days or equivalent doses of other steroids are allowed).

6. Other malignancies within the past 5 years, except for radically treated cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, breast carcinoma in situ, and cervical carcinoma in situ.

7. Systemic anti-tumor therapy within 28 days before starting study treatment, including chemotherapy, immunotherapy, biological therapy (tumor vaccine, cytokines, or growth factors to control cancer), etc.

8. Major surgery within 28 days or radiation therapy within 90 days prior to starting study treatment.

9. Anti-cancer Chinese herbal medicine or Chinese patent medicine within 7 days prior to starting study treatment.

10. Administration of live vaccines (except attenuated influenza vaccines) within 28 days prior to starting study treatment.

11. Patients with known history of human immunodeficiency virus infection and/or acquired immunodeficiency syndrome.

12. Patients with active chronic hepatitis B or active hepatitis C. Patients who are positive for hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies at screening must be further tested for hepatitis B virus (HBV) DNA titer (not more than 2500 copies/mL or 1000 IU/mL) and HCV RNA (not more than the lower limit of detection of the assay).

13. Any active infection requiring systemic anti-infective therapy within 14 days prior to starting study treatment.

14. Pregnant or lactating women. 15. Have uncontrolled concomitant disease. 19. Patients with a previous history of mental illness; those who are incapacitated or have limited behavioral ability.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Complete response rate of Sintilimab combined with rituximab followed by R-CHOP regimen | 36 months
  Investigator-assessed complete response rate of Sintilimab combined with rituximab followed by R-CHOP regimen. Complete response ratewas determined on the basis of investigator assessments according to the Lymphoma response to immunomodulatory therapy criteria (LYRIC) for Malignant Lymphoma, 2016. Tumor assessments were performed with CT/MRI with or without PET.Complete response was defined as the disappearance of all evidence of disease, regression of measurable disease, and no new sites.

SECONDARY OUTCOMES:
Objective response rate of Sintilimab combined with rituximab followed by R-CHOP regimen | 36 months
  Investigator-assessed objective response rate of Sintilimab combined with rituximab followed by R-CHOP regimen. The overall response rate (ORR) including complete response (CR), and partial response (PR) was determined on the basis of investigator assessments according to the Lymphoma response to immunomodulatory therapy criteria (LYRIC) for Malignant Lymphoma, 2016. Tumor assessments were performed with CT/MRI with or without PET.
Progression-free survival of whole cohort | 72 months
  Progression-free survival time assessed by investigator for sintilimab combined with rituximab followed by R-CHOP regimen. Statistical analysis will entail descriptive statistics, and survival analysis including Kaplan-Meier estimates, log-rank testing of univariate prognostic factors, Cox proportional hazards analysis, as well as T-testing and regression analysis for comparing continuous variables in correlative study data. PFS was defined as time from diagnosis until relapse or progression, non-protocol re-treatment of lymphoma, or death as a result of any cause.
Duration of response in responding patients | 72 months
  Duration of response to sequential R-CHOP regimen with sintilimab plus rituximab as assessed by the investigator. Duration of response is defined as the time from the date of first occurrence of CR or PR to the date of the first documented PD or death due to any cause.
Overall survival of whole cohort | 72 months
  Overall survival is defined as the time from the treatment date to the death from any cause.
Incidence of Adverse event | 72 months
  Safety of sintilimab combined with rituximab followed by R-CHOP regimen. An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.Adverse events will be graded by the investigator according to the NCI-CTCAE Version 5.0

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun yat-sen university cancer cencer, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data may be shared with the consent of all investigators